CLINICAL TRIAL: NCT07064343
Title: Stand By Me: Anti-Drug Elite Adventure-Based Training Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Katherine Lam, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BDF_ Anti-drug Elite
Record Dates: First submitted 2025-03-27; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2024-11

CONDITIONS: Drug Abuse Prevention
Keywords: Health Promotion; Drug Abusers; The AWARD model; Adventure-based Training Program
MeSH Terms: conditions — Drug Misuse | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): Participants will attend an two day one night adventure-based training program which includes an educational workshop and five adventure-based activities.
  Interventions: Other: Aspirin

INTERVENTIONS:
Other: Aspirin — Participants are required to complete the training program includes an educational workshops and five adventure-based activities. The key educational workshop's topics include: 1) introduction to the drugs, health and legal consequences of drugs especially cocaine, cannabis and ice, 2) anti-drug services, and 3) the AWARD model.
  Other Names: adventure-based training program

SUMMARY:
This project is expected to establish a network of resilient young people with good anti-drug knowledge to mobilize them to assist in current or future anti-drug work, expanding the antidrug capacity of our community. After the project, it is also anticipated that people in this network will continue to assist in the anti-drug work.

DETAILED DESCRIPTION:
In phase 1, the investigators will deliver adventure-based training programs (2-day 1-night camp). Participants will attend in the educational workshop and undergo five adventure-based activities. The key educational workshop's topics include: 1) introduction to the drugs, health and legal consequences of drugs especially cocaine, cannabis and ice, 2) anti-drug services, and 3) the AWARD model.

ELIGIBILITY:
Inclusion Criteria:

1. post-secondary or tertiary education students,
2. aged 18 - 35,
3. able to speak in Cantonese and write in Chinese.

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-09-08 (Estimated); Study Completion 2025-09-08 (Estimated)

PRIMARY OUTCOMES:
BDF Question Set No. 2 | Baseline and 2 days (pre and post intervention)
  To assess knowledge about the harm of drug abuse. Scoring Instruction: Q1 + Q2 + Q3 + Q4 + Q5 + (6-Q6) + Q7 + Q8 + Q9 + Q10. Minimum score: 10 Maximum score: 50.
BDF Question Set No. 24 | baseline and 2 days (pre and post intervention)
  Knowledge about Cannabis-related Harms. Minimum score: 12 Maximum score: 60. total score calculate: Q1 + Q2 + Q3 + Q4 + Q5 + Q6 + Q7+ Q8 + Q9 + Q10 + (6-Q11) + (6-Q12).
BDF Question Set No. 18 | Baseline and 2 days (pre and post intervention)
  To assess permissive attitude towards drug abuse (Secondary school student version). Minimum score: 21 Maximum score: 105. Total scores calculate: Q1 + Q2 + Q3 + Q4 + Q5 + Q6 + Q7 + Q8 + Q9 + Q10 + Q11 + Q12 + Q13 + Q14 + Q15 + Q16 + Q17 + Q18 + Q19 + Q20 + Q21.
BDF Question Set No. 25 | baseline and 2 days (pre and post intervention)
  To assess permissive attitude towards smoking cannabis. Minimum score: 13 Maximum score: 65. Calculate process: Q1 + Q2 + Q3 + Q4 + Q5 + Q6 + Q7+ Q8 + Q9 + Q10 + Q11 + Q12 + Q13.
BDF Question Set No. 26 | Baseline and 2 days (pre and post intervention)
  To assess permissive attitude towards drugs trafficking. Minimum score: 14 Maximum score: 70. Total scores calculate: Q1 + Q2 + (6-Q3) + Q4 + (6-Q5) + Q6 + (6-Q7) + (6-Q8) + Q9 + Q10 + (6-Q11) + Q12 + Q13.
The Chinese version of the 14-item resilience scale | Baseline and 2 days (pre and post intervention)
  The 14-item resilience scale (RS-14) was used to assess the degree of resilience and was a short version of the original resilience scale (RS). The RS-14 was a 14-item and single-factor structure instrument, comprising a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Examples of the items were, "I feel that I can handle many things at a time" and "I keep interested in things". The Chinese translation of the RS-14 was developed with a backtranslation procedure to ensure accuracy. Suitable internal consistency was suggested by a figure of .917 for the coefficient alpha (regarding the RS-14 of the original scale). Further, the original RS-14 was retested after three weeks, and the test-retest reliability of RS-14 was .736 (.595, .837).

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No